CLINICAL TRIAL: NCT06323655
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Three-way Crossover Study in Healthy Subjects to Evaluate the Next-day Residual Effects of 20 mg Tasimelteon
Brief Title: Evaluation of Next-Day Residual Effects of Tasimelteon Compared With Placebo and Active Control in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1201
Record Dates: First submitted 2019-10-18; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tasimelteon (Experimental): single dose
  Interventions: Drug: Tasimelteon; Drug: Active Control Placebo
- Placebo (Placebo Comparator): single dose
  Interventions: Drug: Active Control Placebo; Drug: Tasimelteon Placebo
- Active Control (Active Comparator): single dose
  Interventions: Drug: Tasimelteon Placebo; Drug: Active Control

INTERVENTIONS:
Drug: Tasimelteon — oral capsule
  Arms: Tasimelteon
Drug: Active Control Placebo — oral capsule
  Arms: Placebo; Tasimelteon
Drug: Tasimelteon Placebo — oral capsule
  Arms: Active Control; Placebo
Drug: Active Control — oral capsule
  Arms: Active Control

SUMMARY:
The aim of this study is to investigate next-day residual effects of tasimelteon compared with placebo and active control in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent;
* Healthy subjects with no medical, psychiatric, or current sleep disorders;
* Men and women ages 21 - 55, inclusive;
* Possession of a valid driver's license ≥ 3 years with reported annual mileage ≥ 3,000 km.

Exclusion Criteria:

* Pregnancy or recent pregnancy;
* Subjects who are unable to read or speak English or French.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Next-day effects on simulated driving performance as measured by changes in Standard Deviation of Lateral Position (SDLP) | Day 1 of Treatment Period 1, Treatment Period 2, and Treatment Period 3 (each Period is 1 day, separated by washout)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Laval, Quebec, Canada